CLINICAL TRIAL: NCT00228358
Title: A Phase I Study of Infusion of HER-2/Neu Specific T Cells in Patients With Advanced Stage HER-2/Neu Expressing Cancers Who Have Received a HER-2/Neu Vaccine
Brief Title: Cyclophosphamide or Denileukin Diftitox Followed By Expanding a Patient's Own T Cells in the Laboratory in Treating Patients With HER-2/Neu Overexpressing Metastatic Breast Cancer, Ovarian Cancer, or Non-Small Cell Lung Cancer Previously Treated With HER-2/Neu Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6223; NCI-2009-01547 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2005-09-13; First posted 2005-09-28 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: HER2-positive Breast Cancer; Recurrent Breast Cancer; Recurrent Non-small Cell Lung Cancer; Recurrent Ovarian Epithelial Cancer; Recurrent Ovarian Germ Cell Tumor; Stage IV Breast Cancer; Stage IV Non-small Cell Lung Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Ovarian Germ Cell Tumor
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Ovarian Epithelial | interventions — Cyclophosphamide; denileukin diftitox; Flow Cytometry; Immunoenzyme Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (cellular infusions after cyclophosphamide) (Experimental): Patients receive low-dose cyclophosphamide IV on day -1 and 3 escalating doses of autologous ex vivo-expanded HER2-specific T cells IV over 30 minutes on days 1, 10, and 20.
  Interventions: Drug: ex vivo-expanded HER2-specific T cells; Drug: cyclophosphamide; Other: flow cytometry; Other: immunoenzyme technique
- Group B (cellular infusions after ONTAK conditioning) (Experimental): Patients receive denileukin diftitox IV over 1 hour on day -1 and 3 escalating doses of autologous ex vivo-expanded HER2-specific T cells IV over 30 minutes on days 1, 10, and 20.
  Interventions: Drug: ex vivo-expanded HER2-specific T cells; Biological: denileukin diftitox; Other: flow cytometry; Other: immunoenzyme technique

INTERVENTIONS:
Drug: ex vivo-expanded HER2-specific T cells — Laboratory-expanded T cells, given IV
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Group A (cellular infusions after cyclophosphamide)
Biological: denileukin diftitox — Given IV
  Other Names: DAB389 interleukin-2; DAB389 interleukin-2 immunotoxin; DAB389-IL2; DABIL2
  Arms: Group B (cellular infusions after ONTAK conditioning)
Other: flow cytometry — Intracellular cytokine staining (correlative study)
Other: immunoenzyme technique — ELIspot assay (correlative study)
  Other Names: immunoenzyme techniques

SUMMARY:
This phase I trial studies the safety and the ability to expand laboratory-treated T cells when given together with cyclophosphamide or denileukin diftitox in treating patients with human epidermal growth factor receptor (HER)-2/neu overexpressing metastatic breast cancer, ovarian cancer, or non-small cell lung cancer previously treated with HER-2/neu vaccine. Laboratory-expanded T cells may help the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Biological therapy, such as denileukin diftitox, may stimulate the immune system in different ways and stop tumor cells from growing. Giving laboratory-treated T cells together with cyclophosphamide or denileukin diftitox may allow the immune system to kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility of expanding HER2 specific T cells ex vivo for infusion into subjects who have advanced HER2 overexpressing cancer.

II. To assess the toxicity associated with infusing autologous HER2 specific T cells into patients using either a single dose of cyclophosphamide or ONTAK (denileukin diftitox) prior to T cell infusion.

SECONDARY OBJECTIVES:

I. To investigate to what extent HER2 specific T cell immunity can be boosted in individuals treated with a single dose of cyclophosphamide of ONTAK followed by infusion of autologous HER2 specific T cells.

II. To investigate the potential anti-tumor effects of HER2 specific T cells in patients with HER2 overexpressing advanced-stage cancers.

III. To evaluate how long tumor antigen specific T cell immune augmentation persists in vivo after a single dose of cyclophosphamide or ONTAK followed by infusion of autologous HER2 specific T cells.

OUTLINE: This is a dose-escalation study of ex vivo-expanded HER2-specific T cells. Patients are assigned to 1 of 2 treatment groups.

GROUP A: Patients receive low-dose cyclophosphamide intravenously (IV) on day -1 and 3 escalating doses of autologous ex vivo-expanded HER2-specific T cells IV over 30 minutes on days 1, 10, and 20.

GROUP B: Patients receive ONTAK (denileukin diftitox) IV over 1 hour on day -1 and 3 escalating doses of autologous ex vivo-expanded HER2-specific T cells IV over 30 minutes on days 1, 10, and 20.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients with progressive HER2/neu overexpressing metastatic breast, ovarian, or non-small cell lung cancer not considered curable by conventional therapies, including trastuzumab

  * Extra-skeletal disease that can be accurately measured >= 10 mm by standard imaging techniques that can include but not limited to computed tomography (CT), positron emission tomography (PET), magnetic resonance imaging (MRI)
  * Skeletal or bone-only disease which is measurable by Fludeoxyglucose F 18 (FDG) PET imaging will also be allowed
  * Patients with ovarian cancer may have measurable disease; however, their only indication of progression may be an abnormal CA-125
* Patients must have documented HER-2/neu overexpression in their tumor (either primary or metastasis) as was required per the eligibility criteria of their original vaccination protocol
* Patients must have received HER2-specific vaccinations while enrolled on a HER2 vaccine protocol approved at the University of Washington Human Subjects Division
* Patients must have undergone leukapheresis after vaccination through a protocol approved at the University of Washington Human Subjects Division and have product stored for clinical use
* Subjects must have a Performance Status Score (Zubrod/Eastern Cooperative Oncology Group [ECOG] Scale) = 0 or 1
* Patients can be currently receiving trastuzumab and/or lapatinib and/or hormonal therapy and/or bisphosphonate therapy

  * Patients on trastuzumab and/or lapatinib must have adequate cardiac function as demonstrated by multi gated acquisition (MUGA) scan or echocardiogram (ECHO) within 90 days of eligibility determination
* Patients must be off all immunosuppressive treatments, and/or systemic steroid therapy, for at least 14 days prior to initiation of study treatment
* Patients must be off chemotherapy and trastuzumab for at least 1 week prior to the first infusion of T cells
* Men and women of reproductive ability must agree to contraceptive use during the study and for one month after the final T cell infusion
* Patients with a history of brain metastases must have a stable head imaging study within 30 days of enrollment
* White blood cells (WBC) >= 3000/mm^3
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Hemoglobin (Hgb) >= 10 mg/dl
* Platelets >= 75,000mm^3
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min
* Total bilirubin =< 2.5 mg/dl
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 3 times ULN

Exclusion Criteria:

* Concurrent enrollment in other treatment studies
* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy
  * Unstable angina within the last 4 months prior to enrollment
  * New York Heart Association functional class III-IV heart failure on active treatment
* Patients with any clinically significant autoimmune disease uncontrolled with treatment
* Pregnant or breast-feeding women
* Known history of hypersensitivity to diphtheria toxin or interleukin (IL)-2 (only for subjects enrolled in Group B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-06; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Feasibility of expanding HER2 specific T cells ex vivo to achieve a target T cell expansion of 1x10^10 HER2 specific T cells | Up to day 40
  The procedure will be defined as feasible if the minimum target expansion of HER2 specific T cells is achieved in 2/3 expansions in 4/5 subjects within an arm.
Safety of infusing HER2 specific T cells | Up to day 40
  Toxicity grading will be evaluated according to the CTEP CTCAE v3.0 criteria. A specific dose of HER2 specific T cells will be defined as safe if 4 of 5 subjects in a study arm tolerate that dose without dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Number of patients in whom the precursor frequency of antigen specific T cells is increased by 10-fold over baseline within one week after the last infusion | Up to one week following last infusion
Number of patients in whom an immune response is demonstrated if baseline immune response was below detection | Up to one week following last infusion
HER2 specific CD4+ or CD8+ precursor frequencies as assessed by cytokine flow cytometry or ELISPOT | Up to 1 year following last infusion
Anti-tumor effects of HER2 specific T cells as assessed by RECIST criteria | Day 40
Persistence of T cell immune augmentation in vivo after adoptive transfer of HER2 specific T cells | Up to 1 year following last infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States